CLINICAL TRIAL: NCT02844023
Title: Biomarkers in Giant Cells Arteritis
Acronym: BioACG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment failure
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC15.198
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Giant Cells Arteritis
Keywords: Arteritis; Biomarker; Horton disease
MeSH Terms: conditions — Arteritis; Giant Cell Arteritis | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient with giant gells arteritis (Other): 50 patients with giant gells arteritis
  Interventions: Behavioral: Clinical evaluation; Other: Paraclinical evaluation; Device: Imaging; Other: Ophthalmologic examination
- Control patients (Other): 50 control patients : blood from French national blood service (EFS)
  Interventions: Biological: Dosage of biomarkers

INTERVENTIONS:
Behavioral: Clinical evaluation — With questionnaire.
  Arms: Patient with giant gells arteritis
Other: Paraclinical evaluation — Symptom inflammatory, biomarkers.
  Arms: Patient with giant gells arteritis
Device: Imaging — Thoraco-abdominal scanner injected or PET scanner if contraindication for scanner.
  Arms: Patient with giant gells arteritis
Other: Ophthalmologic examination
  Arms: Patient with giant gells arteritis
Biological: Dosage of biomarkers — Control patients.
  Arms: Control patients

SUMMARY:
Giant cells arteritis or Horton disease is a vasculitis that affects great vessels. This is the most frequent vasculitis of the population over the age of 50. This vasculitis is at the origin of an inflammatory infiltrate of arterial tunics, essentially composed of lymphocytes. Clinical signs are a deterioration of general state, unusual cephalgias, jaw pain, scalp hyperesthesia, but can also be serious ischemic complication, especially ophthalmologic with the possibility to go blind. Until now, the standard treatment is a high dosage corticosteroid therapy.

Diagnosis is based on criterias of the American College of Rheumatology, dating back to 1990. The relapse rate is important, ranging from 10 to 64 % according to studies. There are also issues of becoming dependent on steroid.

So it is important to determine new diagnosis markers and a therapeutic following of giant cells arteritis.

With this study several biomarkers of inflammation will be studied in order to determine if one ore many of them have a good sensitivity and special feature for diagnosis and following of giant cells arteritis.

The main goal is to determine a new diagnosis marker for giant cells arteritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from giant cells arteritis.
* Inclusion while discovery of symptoms, or during relapse.

Exclusion Criteria:

* Healthy volunteer
* Treatment with corticosteroid since more than 8 days for a patient suffering from giant cells arteritis, exept for patients under corticosteroid for a polymyalgia rheumatica.
* Other diseases than giant cells arteritis that could introduce an inflammatory symptom, especially a tumoral process in progress or a chronic inflammatory disease (any other one than giant cells arteritis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Biomarkers's serum sampling | 3 minutes
  For dosage of biomarkers in serum, like serum amyloid A or interleukins.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Bouillet, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Hachulla E, Boivin V, Pasturel-Michon U, Fauchais AL, Bouroz-Joly J, Perez-Cousin M, Hatron PY, Devulder B. Prognostic factors and long-term evolution in a cohort of 133 patients with giant cell arteritis. Clin Exp Rheumatol. 2001 Mar-Apr;19(2):171-6. PMID 11326479
- [Background] Graham E, Holland A, Avery A, Russell RW. Prognosis in giant-cell arteritis. Br Med J (Clin Res Ed). 1981 Jan 24;282(6260):269-71. doi: 10.1136/bmj.282.6260.269. PMID 6779980
- [Background] Alba MA, Garcia-Martinez A, Prieto-Gonzalez S, Tavera-Bahillo I, Corbera-Bellalta M, Planas-Rigol E, Espigol-Frigole G, Butjosa M, Hernandez-Rodriguez J, Cid MC. Relapses in patients with giant cell arteritis: prevalence, characteristics, and associated clinical findings in a longitudinally followed cohort of 106 patients. Medicine (Baltimore). 2014 Jul;93(5):194-201. doi: 10.1097/MD.0000000000000033. PMID 25181312
- [Background] Proven A, Gabriel SE, Orces C, O'Fallon WM, Hunder GG. Glucocorticoid therapy in giant cell arteritis: duration and adverse outcomes. Arthritis Rheum. 2003 Oct 15;49(5):703-8. doi: 10.1002/art.11388. PMID 14558057
- [Background] Maffioli L, Mazzone A. Giant-cell arteritis and polymyalgia rheumatica. N Engl J Med. 2014 Oct 23;371(17):1652-3. doi: 10.1056/NEJMc1409206. No abstract available. PMID 25337761
- [Background] Kermani TA, Schmidt J, Crowson CS, Ytterberg SR, Hunder GG, Matteson EL, Warrington KJ. Utility of erythrocyte sedimentation rate and C-reactive protein for the diagnosis of giant cell arteritis. Semin Arthritis Rheum. 2012 Jun;41(6):866-71. doi: 10.1016/j.semarthrit.2011.10.005. Epub 2011 Nov 25. PMID 22119103
- [Background] Laria A, Zoli A, Bocci M, Castri F, Federico F, Ferraccioli GF. Systematic review of the literature and a case report informing biopsy-proven giant cell arteritis (GCA) with normal C-reactive protein. Clin Rheumatol. 2012 Sep;31(9):1389-93. doi: 10.1007/s10067-012-2031-3. Epub 2012 Jul 22. PMID 22820967
- [Background] Yoeruek E, Szurman P, Tatar O, Weckerle P, Wilhelm H. Anterior ischemic optic neuropathy due to giant cell arteritis with normal inflammatory markers. Graefes Arch Clin Exp Ophthalmol. 2008 Jun;246(6):913-5. doi: 10.1007/s00417-007-0762-7. Epub 2008 Apr 2. PMID 18386041
- [Background] Kyle V, Cawston TE, Hazleman BL. Erythrocyte sedimentation rate and C reactive protein in the assessment of polymyalgia rheumatica/giant cell arteritis on presentation and during follow up. Ann Rheum Dis. 1989 Aug;48(8):667-71. doi: 10.1136/ard.48.8.667. PMID 2782977
- [Background] Kieffer P, Hinschberger O, Ciobanu E, Jaeger-Bizet F, Drabo A, Mostoufizadeh T, Martzolff L. [Clinical and biological efficacy of tocilizumab in giant cell arteritis: report of three patients and literature review]. Rev Med Interne. 2014 Jan;35(1):56-9. doi: 10.1016/j.revmed.2012.12.012. Epub 2013 Sep 26. French. PMID 24075627
- [Background] Salvarani C, Magnani L, Catanoso M, Pipitone N, Versari A, Dardani L, Pulsatelli L, Meliconi R, Boiardi L. Tocilizumab: a novel therapy for patients with large-vessel vasculitis. Rheumatology (Oxford). 2012 Jan;51(1):151-6. doi: 10.1093/rheumatology/ker296. Epub 2011 Nov 10. PMID 22075063
- [Background] Unizony S, Arias-Urdaneta L, Miloslavsky E, Arvikar S, Khosroshahi A, Keroack B, Stone JR, Stone JH. Tocilizumab for the treatment of large-vessel vasculitis (giant cell arteritis, Takayasu arteritis) and polymyalgia rheumatica. Arthritis Care Res (Hoboken). 2012 Nov;64(11):1720-9. doi: 10.1002/acr.21750. PMID 22674883
- [Background] Samson M, Bonnotte B. [Giant-cell arteritis pathogenesis]. Presse Med. 2012 Oct;41(10):937-47. doi: 10.1016/j.lpm.2012.07.005. Epub 2012 Aug 14. French. PMID 22902103
- [Background] Martinez-Taboada VM, Alvarez L, RuizSoto M, Marin-Vidalled MJ, Lopez-Hoyos M. Giant cell arteritis and polymyalgia rheumatica: role of cytokines in the pathogenesis and implications for treatment. Cytokine. 2008 Nov;44(2):207-20. doi: 10.1016/j.cyto.2008.09.004. Epub 2008 Nov 4. PMID 18986814
- [Background] Ly KH, Liozon E, Fauchais AL, Vidal E. [Pathophysiology of giant cell arteritis]. Rev Med Interne. 2013 Jul;34(7):392-402. doi: 10.1016/j.revmed.2013.02.037. Epub 2013 Mar 23. French. PMID 23528439
- [Background] Ly KH, Regent A, Tamby MC, Mouthon L. Pathogenesis of giant cell arteritis: More than just an inflammatory condition? Autoimmun Rev. 2010 Aug;9(10):635-45. doi: 10.1016/j.autrev.2010.05.002. Epub 2010 May 8. PMID 20457278
- [Background] Weyand CM, Younge BR, Goronzy JJ. IFN-gamma and IL-17: the two faces of T-cell pathology in giant cell arteritis. Curr Opin Rheumatol. 2011 Jan;23(1):43-9. doi: 10.1097/BOR.0b013e32833ee946. PMID 20827207
- [Background] Visvanathan S, Rahman MU, Hoffman GS, Xu S, Garcia-Martinez A, Segarra M, Lozano E, Espigol-Frigole G, Hernandez-Rodriguez J, Cid MC. Tissue and serum markers of inflammation during the follow-up of patients with giant-cell arteritis--a prospective longitudinal study. Rheumatology (Oxford). 2011 Nov;50(11):2061-70. doi: 10.1093/rheumatology/ker163. Epub 2011 Aug 25. PMID 21873264
- [Background] Garcia-Martinez A, Hernandez-Rodriguez J, Espigol-Frigole G, Prieto-Gonzalez S, Butjosa M, Segarra M, Lozano E, Cid MC. Clinical relevance of persistently elevated circulating cytokines (tumor necrosis factor alpha and interleukin-6) in the long-term followup of patients with giant cell arteritis. Arthritis Care Res (Hoboken). 2010 Jun;62(6):835-41. doi: 10.1002/acr.20043. PMID 20535794
- [Background] Ma-Krupa W, Jeon MS, Spoerl S, Tedder TF, Goronzy JJ, Weyand CM. Activation of arterial wall dendritic cells and breakdown of self-tolerance in giant cell arteritis. J Exp Med. 2004 Jan 19;199(2):173-83. doi: 10.1084/jem.20030850. PMID 14734523
- [Background] Samson M, Audia S, Martin L, Janikashvili N, Bonnotte B. Pathogenesis of giant cell arteritis: new insight into the implication of CD161+ T cells. Clin Exp Rheumatol. 2013 Jan-Feb;31(1 Suppl 75):S65-73. Epub 2013 Apr 19. PMID 23663684
- [Background] Samson M, Audia S, Fraszczak J, Trad M, Ornetti P, Lakomy D, Ciudad M, Leguy V, Berthier S, Vinit J, Manckoundia P, Maillefert JF, Besancenot JF, Aho-Glele S, Olsson NO, Lorcerie B, Guillevin L, Mouthon L, Saas P, Bateman A, Martin L, Janikashvili N, Larmonier N, Bonnotte B. Th1 and Th17 lymphocytes expressing CD161 are implicated in giant cell arteritis and polymyalgia rheumatica pathogenesis. Arthritis Rheum. 2012 Nov;64(11):3788-98. doi: 10.1002/art.34647. PMID 22833233
- [Background] Lachmann HJ, Goodman HJ, Gilbertson JA, Gallimore JR, Sabin CA, Gillmore JD, Hawkins PN. Natural history and outcome in systemic AA amyloidosis. N Engl J Med. 2007 Jun 7;356(23):2361-71. doi: 10.1056/NEJMoa070265. PMID 17554117
- [Background] Hachulla E, Saile R, Parra HJ, Hatron PY, Gosset D, Fruchart JC, Devulder B. Serum amyloid A concentrations in giant-cell arteritis and polymyalgia rheumatica: a useful test in the management of the disease. Clin Exp Rheumatol. 1991 Mar-Apr;9(2):157-63. PMID 1711943
- [Background] Blume JD. Bounding Sample Size Projections for the Area Under a ROC Curve. J Stat Plan Inference. 2009 Mar 1;139(1):711-721. doi: 10.1016/j.jspi.2007.09.015. PMID 20160839